CLINICAL TRIAL: NCT02186015
Title: Safety, Feasibility and Efficacy of Vitamin D Supplementation in Women With Metastatic Breast Cancer (SAFE-D)
Acronym: SAFE-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Patricia Sheean, Research Associate, Loyola University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206519
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Adult Women; Metastatic Breast Cancer; Estrogen Receptor Positive
Keywords: Metastatic Breast Cancer; MBC; Vitamin D Supplementation; Symptom Management
MeSH Terms: conditions — Breast Neoplasms | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Experimental): All participants will receive 50,000 IU weekly supplementation of cholecalciferol for 8 weeks.
  Interventions: Drug: Cholecalciferol
- Vitamin D sufficient (No Intervention): All participants were ineligible for the intervention due to sufficient serum 25(OH)D levels at screening/baseline.

INTERVENTIONS:
Drug: Cholecalciferol — Enrolled women will receive 50,000 IU weekly supplementation of cholecalciferol for 8 weeks.
  Other Names: Vitamin D3; Vitamin D
  Arms: Cholecalciferol

SUMMARY:
Background: Several clinical trials are underway to investigate if variable forms of vitamin D (D2 vs. D3) prescribed at different doses (10,000-50,000 IUs/week) can improve the side-effects associated with treatment for estrogen receptor positive (ER+) breast cancer, specifically aromatase inhibitors (AIs.) Presumably for generalizability and potential safety purposes, these trials predominantly exclude women with metastatic breast cancer (MBC); a rapidly expanding sector of the cancer survivor population who experience significant treatment-related side-effects. Evaluation of the safety of vitamin D3 supplementation is crucial since supplementation can lead to high calcium and importantly, in lab studies have shown that vitamin D3 affects a gene that increases estrogen production. To assure that vitamin D3 does not affect the clinical effects of anti-estrogen therapies, the effect of vitamin D3 supplements on estrogen production requires an evaluation that further explores and defines its potential role in symptom management for this population.

Objectives: This pilot study will evaluate the feasibility of vitamin D3 supplementation in women with MBC, providing much needed data on the preliminary safety and efficacy of this treatment in this patient population. This study will determine: 1) if weekly supplementation of high dose vitamin D3 increases serum vitamin D levels without adverse effects related to such therapy (primary aim); 2) the effects of vitamin D3 supplementation on symptom management (secondary aim); and 3) if vitamin D3 supplementation is associated with improved inflammation (exploratory aim.)

Methods: This is an 8 week "proof of concept" study to monitor laboratory parameters and to assess potential effects on short-term outcomes. Adult, female patients (>=18 years) with ER+ MBC (Stage IV) of any race/ethnicity and a history of vitamin D < 30 mg/dl will be recruited from within and around LUMC. Following current clinical practice guidelines, eligible participants will receive 50,000 IUs of vitamin D3 weekly for 8 weeks. Laboratory values, muscle function and inflammation will be examined pre- and post-supplementation, while symptoms will be assessed at baseline, 4 and 8 weeks post-supplementation. We will assess if increases in vitamin D are associated with clinically significant improvements in symptoms and QOL, and decreased inflammation.

DETAILED DESCRIPTION:
Study Aims

Several clinical trials are underway to investigate if vitamin D2 or D3 provided at various doses (10,000-50,000 IUs/week) can improve the side-effects associated with anti-estrogen therapies, specifically aromatase inhibitors (AIs). However, these current trials use variable forms of vitamin D and predominantly include women with Stage I-III disease, excluding women with metastatic breast cancer. Evaluation of the safety of vitamin D3 supplementation is crucial since supplementation can lead to hypercalcemia and importantly, in vitro studies have shown that vitamin D3 influences the transcription of a gene that increases estrogen production.27,28 To assure that vitamin D3 does not abrogate the clinical effects of anti-estrogen therapies, the effect of vitamin D3 supplementation on estrogen production requires evaluation. Therefore, the overarching goal of this pilot study is to evaluate the safety, feasibility and efficacy of vitamin D3 supplementation in women with MBC. We will address and test the following aims and hypotheses, respectively:

Aim 1: To determine if weekly supplementation of 50,000 IUs of vitamin D3 raises serum levels of 25(OH)D to >30 mg/dl without adverse effects.

Hypothesis 1: Women who are compliant with vitamin D3 supplementation, as evidenced by normalization (>30 mg/dl) or increases in their serum 25(OH)D levels, will not experience significant changes in serum calcium, parathyroid hormone or serum estradiol levels.

Aim 2: To determine the effect of vitamin D3 supplementation on symptom management.

Hypothesis 2: Women who achieve serum concentrations of 25 (OH)D ≥30 mg/dl or experience significant increases in 25(OH)D will exhibit improvements in pain, fatigue, sleep, mood, muscle function and overall quality of life.

Exploratory Aim: To explore the mechanistic effects of vitamin D3 supplementation on inflammatory markers and its potential association with symptom management.

Summary: Evidence from studies involving early stage breast cancer participants confirms that musculoskeletal pain, endocrine related symptoms and mood disturbances are commonly associated with breast cancer treatment, particularly hormone deprivation therapies. The high prevalence of vitamin D deficiency/insufficiency among breast cancer survivors is well accepted and further hypothesized to aggravate treatment-related side effects, particularly arthralgias. Women with MBC are excluded from the majority of on-going vitamin D supplementation trials for safety and generalizability purposes. However, novel therapies are continuing to improve and prolong the lives of these women, resulting in a rapidly expansive group of breast cancer survivors. While vitamin D supplementation is prescribed to correct an underlying nutrient deficiency in the clinical context of preserving bone health, emerging evidence suggests it may have more systemic effects. Thus, vitamin D repletion/supplementation has profound potential implications for women with MBC, whose primary goal of treatment is to minimize the side-effects of treatment in support of optimal quality of life. This study reflects a highly innovative, yet simple therapy that could ultimately provide these survivors with a much needed evidence-based supportive care strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic breast cancer (Stage IV)
2. Histologically confirmed estrogen receptor positive disease
3. Female
4. Serum 25(OH) <30 ng/ml
5. Age ≥ 18 years
6. Pre or post-menopausal
7. ECOG Performance status 0-2
8. Adequate organ function as defined as GFR> 30 mls/min and serum calcium ≤ 10.4 mg/dl
9. Any race/ethnicity
10. English speaking
11. No changes to MBC treatments within 30 days of enrollment and/or deemed clinically stable by their treating physician
12. Willingness to sign a written informed consent and complete questionnaires
13. Cease ingestion of vitamin D supplementation not study related

Exclusion Criteria:

1. Women with Stage I-III breast cancer
2. Serum 25(OH)D levels ≥ 30 ng/ml
3. Untreated CNS involvement
4. History of kidney stones
5. History of renal failure
6. History of hyperparathyroidism
7. History of hypersensitivity to vitamin D
8. Non-English speaking
9. Currently pregnant or lactating, or anticipating pregnancy
10. Unwilling to cease ingestion of calcium supplements (>1000 mg/d)
11. Unwilling or unable to complete informed consent or study questionnaires
12. Psychiatric or other clinical conditions that preclude study compliance
13. Other important medical or safety considerations at the discretion of the investigator and/or study physician, including non-compliance with the study therapy or other activities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03-08 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Sheean, Ph.D., R.D., Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

REFERENCES:
- [Background] Johnson RH, Chien FL, Bleyer A. Incidence of breast cancer with distant involvement among women in the United States, 1976 to 2009. JAMA. 2013 Feb 27;309(8):800-5. doi: 10.1001/jama.2013.776. PMID 23443443
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Reed E, Simmonds P, Haviland J, Corner J. Quality of life and experience of care in women with metastatic breast cancer: a cross-sectional survey. J Pain Symptom Manage. 2012 Apr;43(4):747-58. doi: 10.1016/j.jpainsymman.2011.05.005. Epub 2011 Nov 16. PMID 22088804
- [Background] Goodwin PJ, Ennis M, Pritchard KI, Koo J, Hood N. Prognostic effects of 25-hydroxyvitamin D levels in early breast cancer. J Clin Oncol. 2009 Aug 10;27(23):3757-63. doi: 10.1200/JCO.2008.20.0725. Epub 2009 May 18. PMID 19451439
- [Background] Rose AA, Elser C, Ennis M, Goodwin PJ. Blood levels of vitamin D and early stage breast cancer prognosis: a systematic review and meta-analysis. Breast Cancer Res Treat. 2013 Oct;141(3):331-9. doi: 10.1007/s10549-013-2713-9. Epub 2013 Oct 9. PMID 24104883
- [Background] Napoli N, Vattikuti S, Ma C, Rastelli A, Rayani A, Donepudi R, Asadfard M, Yarramaneni J, Ellis M, Armamento-Villareal R. High prevalence of low vitamin D and musculoskeletal complaints in women with breast cancer. Breast J. 2010 Nov-Dec;16(6):609-16. doi: 10.1111/j.1524-4741.2010.01012.x. PMID 21070438
- [Background] Neuhouser ML, Sorensen B, Hollis BW, Ambs A, Ulrich CM, McTiernan A, Bernstein L, Wayne S, Gilliland F, Baumgartner K, Baumgartner R, Ballard-Barbash R. Vitamin D insufficiency in a multiethnic cohort of breast cancer survivors. Am J Clin Nutr. 2008 Jul;88(1):133-9. doi: 10.1093/ajcn/88.1.133. PMID 18614733
- [Background] Trukova KP, Grutsch J, Lammersfeld C, Liepa G. Prevalence of vitamin D insufficiency among breast cancer survivors. Nutr Clin Pract. 2012 Feb;27(1):122-8. doi: 10.1177/0884533611431461. Epub 2012 Jan 6. PMID 22227726
- [Background] Shao T, Klein P, Grossbard ML. Vitamin D and breast cancer. Oncologist. 2012;17(1):36-45. doi: 10.1634/theoncologist.2011-0278. Epub 2012 Jan 10. PMID 22234628
- [Background] Amir E, Simmons CE, Freedman OC, Dranitsaris G, Cole DE, Vieth R, Ooi WS, Clemons M. A phase 2 trial exploring the effects of high-dose (10,000 IU/day) vitamin D(3) in breast cancer patients with bone metastases. Cancer. 2010 Jan 15;116(2):284-91. doi: 10.1002/cncr.24749. PMID 19918922
- [Background] Simmons C, Amir E, Dranitsaris G, Clemons M, Wong B, Veith R, Cole DE. Altered calcium metabolism in patients on long-term bisphosphonate therapy for metastatic breast cancer. Anticancer Res. 2009 Jul;29(7):2707-11. PMID 19596950
- [Background] Castel LD, Hartmann KE, Mayer IA, Saville BR, Alvarez J, Boomershine CS, Abramson VG, Chakravarthy AB, Friedman DL, Cella DF. Time course of arthralgia among women initiating aromatase inhibitor therapy and a postmenopausal comparison group in a prospective cohort. Cancer. 2013 Jul 1;119(13):2375-82. doi: 10.1002/cncr.28016. Epub 2013 Apr 10. PMID 23575918
- [Background] Niravath P. Aromatase inhibitor-induced arthralgia: a review. Ann Oncol. 2013 Jun;24(6):1443-9. doi: 10.1093/annonc/mdt037. Epub 2013 Mar 6. PMID 23471104
- [Background] Islander U, Jochems C, Lagerquist MK, Forsblad-d'Elia H, Carlsten H. Estrogens in rheumatoid arthritis; the immune system and bone. Mol Cell Endocrinol. 2011 Mar 15;335(1):14-29. doi: 10.1016/j.mce.2010.05.018. Epub 2010 Jun 8. PMID 20685609
- [Background] Din OS, Dodwell D, Wakefield RJ, Coleman RE. Aromatase inhibitor-induced arthralgia in early breast cancer: what do we know and how can we find out more? Breast Cancer Res Treat. 2010 Apr;120(3):525-38. doi: 10.1007/s10549-010-0757-7. Epub 2010 Feb 16. PMID 20157776
- [Background] Soares MJ, Murhadi LL, Kurpad AV, Chan She Ping-Delfos WL, Piers LS. Mechanistic roles for calcium and vitamin D in the regulation of body weight. Obes Rev. 2012 Jul;13(7):592-605. doi: 10.1111/j.1467-789X.2012.00986.x. Epub 2012 Mar 2. PMID 22385576
- [Background] Penckofer S, Kouba J, Byrn M, Estwing Ferrans C. Vitamin D and depression: where is all the sunshine? Issues Ment Health Nurs. 2010 Jun;31(6):385-93. doi: 10.3109/01612840903437657. PMID 20450340
- [Background] Schleithoff SS, Zittermann A, Tenderich G, Berthold HK, Stehle P, Koerfer R. Vitamin D supplementation improves cytokine profiles in patients with congestive heart failure: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2006 Apr;83(4):754-9. doi: 10.1093/ajcn/83.4.754. PMID 16600924
- [Background] Irvin W Jr, Muss HB, Mayer DK. Symptom management in metastatic breast cancer. Oncologist. 2011;16(9):1203-14. doi: 10.1634/theoncologist.2011-0159. Epub 2011 Aug 31. PMID 21880861
- [Background] Eastell R, Adams JE, Coleman RE, Howell A, Hannon RA, Cuzick J, Mackey JR, Beckmann MW, Clack G. Effect of anastrozole on bone mineral density: 5-year results from the anastrozole, tamoxifen, alone or in combination trial 18233230. J Clin Oncol. 2008 Mar 1;26(7):1051-7. doi: 10.1200/JCO.2007.11.0726. PMID 18309940
- [Background] Lonning PE, Geisler J, Krag LE, Erikstein B, Bremnes Y, Hagen AI, Schlichting E, Lien EA, Ofjord ES, Paolini J, Polli A, Massimini G. Effects of exemestane administered for 2 years versus placebo on bone mineral density, bone biomarkers, and plasma lipids in patients with surgically resected early breast cancer. J Clin Oncol. 2005 Aug 1;23(22):5126-37. doi: 10.1200/JCO.2005.07.097. Epub 2005 Jun 27. PMID 15983390
- [Background] Gonnelli S, Cadirni A, Caffarelli C, Petrioli R, Montagnani A, Franci MB, Lucani B, Francini G, Nuti R. Changes in bone turnover and in bone mass in women with breast cancer switched from tamoxifen to exemestane. Bone. 2007 Jan;40(1):205-10. doi: 10.1016/j.bone.2006.06.027. Epub 2006 Aug 14. PMID 16904960
- [Background] Peterson CA, Heffernan ME. Serum tumor necrosis factor-alpha concentrations are negatively correlated with serum 25(OH)D concentrations in healthy women. J Inflamm (Lond). 2008 Jul 24;5:10. doi: 10.1186/1476-9255-5-10. PMID 18652680
- [Background] Giulietti A, van Etten E, Overbergh L, Stoffels K, Bouillon R, Mathieu C. Monocytes from type 2 diabetic patients have a pro-inflammatory profile. 1,25-Dihydroxyvitamin D(3) works as anti-inflammatory. Diabetes Res Clin Pract. 2007 Jul;77(1):47-57. doi: 10.1016/j.diabres.2006.10.007. Epub 2006 Nov 16. PMID 17112620
- [Background] May E, Asadullah K, Zugel U. Immunoregulation through 1,25-dihydroxyvitamin D3 and its analogs. Curr Drug Targets Inflamm Allergy. 2004 Dec;3(4):377-93. doi: 10.2174/1568010042634596. PMID 15584887
- [Background] Krishnan AV, Swami S, Peng L, Wang J, Moreno J, Feldman D. Tissue-selective regulation of aromatase expression by calcitriol: implications for breast cancer therapy. Endocrinology. 2010 Jan;151(1):32-42. doi: 10.1210/en.2009-0855. Epub 2009 Nov 11. PMID 19906814
- [Background] Enjuanes A, Garcia-Giralt N, Supervia A, Nogues X, Mellibovsky L, Carbonell J, Grinberg D, Balcells S, Diez-Perez A. Regulation of CYP19 gene expression in primary human osteoblasts: effects of vitamin D and other treatments. Eur J Endocrinol. 2003 May;148(5):519-26. doi: 10.1530/eje.0.1480519. PMID 12720534
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Wilson IB, Cleary PD. Linking clinical variables with health-related quality of life. A conceptual model of patient outcomes. JAMA. 1995 Jan 4;273(1):59-65. PMID 7996652
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Piper BF, Dibble SL, Dodd MJ, Weiss MC, Slaughter RE, Paul SM. The revised Piper Fatigue Scale: psychometric evaluation in women with breast cancer. Oncol Nurs Forum. 1998 May;25(4):677-84. PMID 9599351
- [Background] Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res. 1997 Jan;42(1):17-41. doi: 10.1016/s0022-3999(96)00216-4. PMID 9055211
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Rantanen T, Era P, Heikkinen E. Maximal isometric strength and mobility among 75-year-old men and women. Age Ageing. 1994 Mar;23(2):132-7. doi: 10.1093/ageing/23.2.132. PMID 8023721
- [Background] Rantanen T, Volpato S, Ferrucci L, Heikkinen E, Fried LP, Guralnik JM. Handgrip strength and cause-specific and total mortality in older disabled women: exploring the mechanism. J Am Geriatr Soc. 2003 May;51(5):636-41. doi: 10.1034/j.1600-0579.2003.00207.x. PMID 12752838
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Carpenter JS, Andrykowski MA. Psychometric evaluation of the Pittsburgh Sleep Quality Index. J Psychosom Res. 1998 Jul;45(1):5-13. doi: 10.1016/s0022-3999(97)00298-5. PMID 9720850
- [Background] Fallowfield LJ, Leaity SK, Howell A, Benson S, Cella D. Assessment of quality of life in women undergoing hormonal therapy for breast cancer: validation of an endocrine symptom subscale for the FACT-B. Breast Cancer Res Treat. 1999 May;55(2):189-99. doi: 10.1023/a:1006263818115. PMID 10481946
- [Background] Cummings SR, Block G, McHenry K, Baron RB. Evaluation of two food frequency methods of measuring dietary calcium intake. Am J Epidemiol. 1987 Nov;126(5):796-802. doi: 10.1093/oxfordjournals.aje.a114716. PMID 3661527
- [Background] Glanz K, Yaroch AL, Dancel M, Saraiya M, Crane LA, Buller DB, Manne S, O'Riordan DL, Heckman CJ, Hay J, Robinson JK. Measures of sun exposure and sun protection practices for behavioral and epidemiologic research. Arch Dermatol. 2008 Feb;144(2):217-22. doi: 10.1001/archdermatol.2007.46. PMID 18283179
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Derived] Maureen Sheean P, Robinson P, Bartolotta MB, Joyce C, Adams W, Penckofer S. Associations Between Cholecalciferol Supplementation and Self-Reported Symptoms Among Women With Metastatic Breast Cancer and Vitamin D Deficiency: A Pilot Study. Oncol Nurs Forum. 2021 May 1;48(3):352-360. doi: 10.1188/21.ONF.352-360. PMID 33856003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a single cancer center and required to be: 1) >18 years of age, 2) English speaking, 3) at a performance status of 0-2, 4) receiving treatment for histologically confirmed ER+ metastatic BC, and 5) clinically stable as judged by their medical oncologist.
Groups:
- No Cholecalciferol: Enrolled women with serum 25 (OH)D greater than or equal to 30 ng/ml received no intervention.
Period: Overall Study
Arm/Group | Cholecalciferol | No Cholecalciferol
Started | 11 | 31
Completed | 10 | 31
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cholecalciferol: Enrolled women with serum 25 (OH)D less than 30 ng/ml received 50,000 IUs weekly supplementation of cholecalciferol for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol | No Cholecalciferol | Total
Number analyzed (Participants) | 11 | 31 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 20 | 30
  >=65 years | 1 | 11 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [46 to 64] | 63 [56 to 70] | 62 [53 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 31 | 42
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 5 | 26 | 31
  Race/Ethnicity: Black | 4 | 0 | 4
  Race/Ethnicity: Hispanic | 2 | 4 | 6
  Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Midwest United States
  Participants
    United States | 11 | 31 | 42
Employment status [Count of Participants; unit: Participants]
  Paid full- or part-time work | 6 | 12 | 18
  Retired without disability | 1 | 12 | 13
  Retired with disability | 2 | 6 | 8
  Unemployed | 2 | 1 | 3
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.3 [25.3 to 40.1] | 27.8 [23.7 to 33.2] | 27.5 [24.1 to 33.2]
Stage IV at diagnosis [Count of Participants; unit: Participants] — Metastatic breast cancer at diagnosis
  Participants
    Yes | 4 | 8 | 12
    No | 7 | 23 | 30
Duration of metastatic breast cancer [Median (Inter-Quartile Range); unit: months] | 7 [3 to 14] | 19 [5 to 45] | 13 [5 to 33]
Metastatic sites [Count of Participants; unit: Participants]
  1 or 2 | 9 | 25 | 34
  Greater than 2 | 2 | 6 | 8
Eastern Cooperative Oncology Group [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance status describes patients' level of functioning, where higher scores indicate lower levels of functioning.
  Participants
    0 | 5 | 11 | 16
    1 | 6 | 19 | 25
    2 | 0 | 1 | 1
Radiation therapy for metastates [Count of Participants; unit: Participants]
  Yes | 3 | 10 | 13
  No | 8 | 21 | 29
Surgery for breast cancer [Count of Participants; unit: Participants]
  None | 6 | 5 | 11
  Lumpectomy | 4 | 14 | 18
  Mastectomy | 1 | 12 | 13
Serum 25(OH)D [Median (Inter-Quartile Range); unit: ng/ml] | 17 [13 to 26] | 38 [34 to 44] | 34 [29 to 42]

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum 25(OH)D
Description: Change in laboratory serum value of 25(OH)D at 8 weeks post-supplementation for participants who received weekly supplementation of 50,000 IUs of vitamin D3. Change is expressed as laboratory serum value of 25(OH)D at 8 weeks minus baseline. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did not have laboratory serum value of 25(OH)D at week 8. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Cholecalciferol: Enrolled women received 50,000 IUs weekly supplementation of cholecalciferol for 8 weeks.
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
ng/ml | 32 [22 to 40] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in serum 25(OH)D from week 0 to week 8; Test type: Superiority — A Wilcoxon signed rank test was performed; p < 0.01, Wilcoxon signed rank test

2. Secondary Outcome: Change in Worst Pain Rating From the Beck Pain Scale
Description: Assessment of pain using the Beck Pain Scale at weeks 0 and 8. This is a Likert scale item where a score of 0 corresponds to no pain and a score of 10 corresponds to worst pain. Change is calculated as the worst pain rating at 8 weeks minus the worst pain rating at 0 weeks.Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
score on a scale | 0 [-3 to 0] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in worst pain rating from week 0 to week 8; Test type: Superiority — A Wilcoxon signed rank test was performed; p = 0.24, Wilcoxon signed rank test

3. Secondary Outcome: Change in Fatigue
Description: Assessment of fatigue using the Piper Fatigue Scale at weeks 0 and 8. The Piper Fatigue Scale is the average of 22 numeric items, with higher scores indicating greater fatigue [range of scores: 0-10]. Change is calculated as the fatigue score at 8 weeks minus fatigue score at 0 weeks. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did not have assessment of fatigue at week 8. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
units on a scale | -0.5 [-1.7 to 0.1] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in fatigue score from week 0 to week 8; Test type: Superiority; p = 0.09, Wilcoxon signed rank test

4. Secondary Outcome: Change in Mood
Description: Assessment of mood using the Patient Health Questionnaire 8 (PHQ-8) at weeks 0 and 8. The PHQ-8 ranges from 0-24 with higher scores indicating more distress. Change was assessed as PHQ-8 score at 8 weeks minus 0 weeks. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did not have assessment of mood at 8 weeks. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
score on a scale | -1 [-4 to 2] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in mood score from week 0 to week 8; Test type: Superiority; p = 0.17, Wilcoxon signed rank test

5. Secondary Outcome: Change in Muscle Function
Description: Assessment of muscle function using a hand dynamometer at weeks 0 and 8. Change in dominant handgrip strength in kilograms was calculated as 8 weeks minus 0 weeks. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did not have hand dynamometer data at 8 weeks. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
kilograms | -0.2 [-1.0 to 7.3] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in dominant handgrip strength from week 0 to week 8; Test type: Superiority; p = 0.50, Wilcoxon signed rank test

6. Secondary Outcome: Change in Sleep Quality Assessment
Description: Assessment of sleep using the Pittsburgh Sleep Quality Index (PSQI) at weeks 0 and 8. Scores range from 0-21 with higher scores indicating poorer sleep quality. Change was calculated as week 8 minus week 0 PSQI. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did report the Pittsburgh Sleep Quality Index at week 8. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
score on a scale | -1 [-4 to 4] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in sleep quality assessment from week 0 to week 8; Test type: Superiority; p = 0.16, Wilcoxon signed rank test

7. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-breast
Description: Assessment of quality of life using the functional assessment of cancer therapy-breast symptoms at weeks 0 and 8. Scores range from 0-40 with higher scores indicating better quality of life.
  Change was calculated as week 8 score minus week 0 score. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did not have the Functional assessment of cancer therapy-breast at 8 weeks. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
score on a scale | 0 [-7 to 17] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in functional assessment of cancer therapy-breast score from week 0 to week 8; Test type: Superiority; p = 0.75, Wilcoxon signed rank test

8. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-endocrine
Description: Assessment of quality of life using the functional assessment of cancer therapy- endocrine symptoms at weeks 0 and 8. Scores range from 0-76 with higher scores indicating better quality of life. Change was not assessed for participants in the 'no cholecalciferol' arm since they did not receive weekly supplementation and were not followed over time.
Time Frame: 0, 8 weeks
Population: 1 participant who initiated supplementation of cholecalciferol did not have the Functional assessment of cancer therapy-endocrine at 8 weeks. Follow up laboratory and/or questionnaire data were not collected for women in the 'no cholecalciferol' arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cholecalciferol | No Cholecalciferol
Number analyzed (Participants) | 10 | 0
score on a scale | 9 [-2 to 14] |
Statistical Analysis 1: Comparison: Cholecalciferol; The null hypothesis is that there is 0 change in functional assessment of cancer therapy-endocrine score from week 0 to week 8; Test type: Superiority; p = 0.19, Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Intervention: Enrolled women with serum 25 (OH)D less than 30 ng/ml received 50,000 IUs weekly supplementation of cholecalciferol for 8 weeks
- No Intervention: Enrolled women without serum 25 (OH)D greater than or equal to 30 ng/ml received no intervention.
Arm/Group | Intervention | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/31
Other Adverse Events (participants affected / at risk) | 3/11 | 0/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=11) | No Intervention (N=31)
Nausea (Gastrointestinal disorders) | 3 (3) | 0
Upper respiratory infection (Infections and infestations) | 2 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2014-11-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02186015/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02186015/SAP_001.pdf
  • Informed Consent Form (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT02186015/ICF_002.pdf